CLINICAL TRIAL: NCT05650411
Title: ULTRATHIN-STRUT BIODEGRADABLE POLYMER SIROLIMUS-ELUTING STENTS COMBINED WITH P2Y12 INHIBITOR-BASED SINGLE ANTIPLATELET THERAPY AFTER A SHORT DUAL ANTIPLATELET THERAPY REGIMEN VERSUS CONVENTIONAL DUAL ANTIPLATELET THERAPY FOR UNPROTECTED LEFT MAIN CORONARY ARTERY DISEASE
Brief Title: Ultrathin-strut Biodegradable Polymer Sirolimus-eluting Stents With P2Y12 Inhibitor-based Single Antiplatelet Therapy vs. Conventional DAPT for Unprotected Left Main Coronary Artery Disease (ULTIMATE-LM)
Acronym: ULTIMATE-LM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IGLESIAS Juan Fernando (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, IGLESIAS Juan Fernando, MD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1204
Record Dates: First submitted 2022-12-04; First posted 2022-12-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Left Main Coronary Artery Stenosis
Keywords: P2Y12 inhibitor-based single antiplatelet therapy; Dual antiplatelet therapy; Left main coronary artery disease; Percutaneous coronary intervention; Ultrathin-strut; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P2Y12 inhibitor-based single antiplatelet therapy after a short DAPT strategy arm (Experimental): Successful LMCA PCI with ≥1 Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India).
  P2Y12 inhibitor SAPT with any of the commercially available oral P2Y12 inhibitors (ticagrelor, or prasugrel 10 mg) after a short DAPT course during 2 years after the index LMCA procedure.
  At the discretion of the investigator, aspirin will be discontinued after LMCA PCI, or continued during the hospital stay. In all cases, aspirin will be discontinued at latest at hospital discharge.
  Interventions: Device: LMCA PCI with Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India).; Drug: P2Y12 inhibitor-based SAPT after short DAPT
- Conventional DAPT strategy arm (Active Comparator): Successful LMCA PCI with ≥1 Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India).
  DAPT combining aspirin and any of the commercially available oral P2Y12 receptor inhibitors (clopidogrel, ticagrelor, or prasugrel) during 6 or 12 months followed by aspirin-based SAPT.
  In patients with index ACS presentation and who have tolerated DAPT for 12 months without bleeding complications, a prolonged DAPT course with aspirin and ticagrelor 60 mg bd (clopidogrel or prasugrel allowed, if patient not eligible for treatment with ticagrelor) beyond 12 months may be considered in those patients with high thrombotic risk and without an increased risk for major or life-threatening bleeding, and those with moderately elevated thrombotic risk.
  Interventions: Device: LMCA PCI with Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India).; Drug: Conventional DAPT

INTERVENTIONS:
Device: LMCA PCI with Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India). — Successful LMCA PCI with ≥1 Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India).
Drug: P2Y12 inhibitor-based SAPT after short DAPT — Potent P2Y12 inhibitor-based SAPT (ticagrelor 90 mg bd, or prasugrel 5 or 10 mg od, at the discretion of the investigator) during 2 years. Aspirin stopped after LMCA or at latest at hospital discharge.
  Arms: P2Y12 inhibitor-based single antiplatelet therapy after a short DAPT strategy arm
Drug: Conventional DAPT — 6 to 12 months of DAPT combining aspirin (≥75 mg od) and a P2Y12 inhibitor (clopidogrel 75 mg od, ticagrelor 90 mg bd, prasugrel 5 or 10 mg od at the discretion of the investigator) followed by aspirin SAPT.
  Arms: Conventional DAPT strategy arm

SUMMARY:
The management of patients with unprotected left main coronary artery (LMCA) disease undergoing percutaneous coronary intervention (PCI) in contemporary interventional cardiology practice remains matter of intense debate. Particularly, the combination of the optimal drug-eluting stent (DES) selection and antiplatelet regimen for patients who require LMCA PCI remains undetermined.

Newer-generation drug-eluting stents with ultrathin-strut metallic platforms have been shown to reduce the risk of target lesion failure compared with thicker-strut drug-eluting stents among all-comer patients undergoing PCI, a difference mainly driven by a lower risk of ischemia-driven target lesion revascularization. In the TALENT prospective, single-blind, multicenter, randomized controlled trial that included 1'435 all-comer patients undergoing PCI, the Supraflex ultrathin-strut biodegradable polymer sirolimus-eluting stent was found non-inferior to the Xience® thin-strut permanent polymer everolimus-eluting stent (Abbott Vascular, USA) with regards to the device-oriented composite clinical endpoint (DoCE), a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization, at 12 months of follow-up. However, the TALENT trial included only 31 (1.5%) lesions located in the left main coronary artery. In the COMPARE 60/80 HBR investigator-initiated, multicenter, prospective randomized trial which included a total of 732 patients at high-bleeding risk undergoing PCI with the Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent or the Ultimaster Tansei (Terumo Corp., Tokyo, Japan), the rates of the primary endpoint of the net adverse clinical endpoint, defined as a composite of cardiac death, myocardial infarction, target vessel revascularization, stroke, or BARC 3 or 5 major bleeding events at 12 months were similar in the Supraflex Cruz and the Ultimaster Tansei groups, meeting the prespecified criterion for non-inferiority of the Supraflex Cruz DES compared to the Ultimaster Tansei DES. The safety and efficacy of the Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent combined with potent P2Y12 inhibitor aspirin-free SAPT among all-comer patients undergoing PCI for complex coronary lesions, such as patients with LMCA stenosis, have however not been investigated to date.

Recent evidence from a large-scale meta-analysis of several randomized clinical trials including >32'000 patients indicated that 1-3 months of DAPT followed by P2Y12 inhibitor single antiplatelet therapy (SAPT) after second-generation DES implantation was associated with lower risk for major bleeding and similar risk for adverse ischemic outcomes compared with conventional DAPT. These findings suggest that P2Y12 inhibitor SAPT following a short DAPT course (1-3 months) may represent a valuable treatment option for patients undergoing PCI with newer-generation DES compared to standard conventional 12 months DAPT, but this strategy has never been investigated in dedicated randomized clinical trials focused on patients at highest-risk for ischaemic events, such as patients undergoing LMCA PCI.

The ULTIMATE-LM randomized trial aims at filling this current gap of knowledge, which may have large impact on clinical practice and international guidelines. ULTIMATE-LM will be the first randomized clinical trial to investigate the safety and efficacy of a novel ultrathin-strut biodegradable polymer drug-eluting stent (Supraflex Cruz, Sahajanand Medical Technologies Ltd., Surat, India)) combined with P2Y12 inhibitor-based single antiplatelet therapy among patients undergoing PCI for LMCA disease.

DETAILED DESCRIPTION:
1. Myocardial revascularization for left main coronary artery disease

   Significant left main coronary artery disease (LMCA) is observed in 5-7% of patients undergoing coronary angiography. Coronary revascularization for patients with LMCA disease with stenosis >50% and documented ischemia or FFR ≤0.80 for diameter stenosis <90%, is recommended with a class of recommendation I and level of evidence (LOE) A by the 2018 European Society of Cardiology (ESC) guidelines for myocardial revascularization. However, the optimal management of patients with LMCA disease requiring myocardial revascularization in contemporary clinical practice remains matter of debate.
2. Coronary artery bypass grafting vs. percutaneous coronary intervention for left main coronary artery disease

   The available evidence from randomized controlled trials (RCTs) and meta-analyses comparing coronary artery bypass grafting (CABG) with percutaneous coronary intervention (PCI) using drug-eluting stents (DESs) among patients with LMCA suggests equivalent results for the safety composite of death, myocardial infarction (MI), and stroke up to 5 years of follow-up. A significant interaction with time is notable, providing early benefit for PCI in terms of MI and peri-interventional stroke, which is subsequently offset by a higher risk of spontaneous MI during long-term follow-up. The need for repeat revascularization is higher with PCI than with CABG. The largest RCT among patients with LMCA disease so far performed, EXCEL (Evaluation of XIENCE versus Coronary Artery Bypass Surgery for Effectiveness of Left Main Revascularization), compared CABG with PCI using new-generation DESs among 1,905 patients with significant LMCA. At 3 years of follow-up, the primary endpoint of death, stroke, or MI occurred with similar frequency in the CABG and PCI group (14.7% vs. 15.4%; HR 1.00, 95% CI 0.79-1.26, p=0.98). The pre-planned landmark analysis from 30 days to 3 years showed a significant difference for the primary endpoint in favour of CABG (7.9% vs. 11.5%, p=0.02). The NOBLE (Nordic-Baltic-British Left Main Revascularization Study) randomized trial compared CABG with PCI using new-generation biolimus-eluting stents among 1,201 patients with significant LM disease (mean SYNTAX score of 23). At a median follow-up of 3.1 years, the primary endpoint of death, non-procedural MI, stroke, and repeat revascularization occurred more frequently in the PCI than the CABG group (29% vs. 19%; HR 1.48, 95% CI 1.11-1.96, p=0.007). A recent collaborative individual patient data pooled analysis of RCTs including 11,518 patients reviewed the currently available evidence from RCTs comparing CABG with PCI for LMCA or multivessel disease. The primary outcome was all-cause mortality. In the overall cohort, CABG was associated with a significant survival benefit during a mean follow-up of 3.8±1.4 years (5-year all-cause mortality 11.2% after PCI vs. 9.2% after CABG; HR 1.20, 95% CI 1.06-1.37, p=0.0038). There was a linear trend for HRs of death increasing with increasing SYNTAX terciles (p=0.0011 for trend). However, among 4,478 patients with LMCA, those randomly assigned to CABG or PCI with a mean follow-up of 3.4±1.4 years reported similar risks for the primary outcome all-cause mortality (PCI, 10.7% vs. CABG, 10.5%; HR 1.07, 95% CI 0.87-1.33, p=0.52) at 5 years. There were no significant differences in mortality between PCI and CABG in subgroup analyses according to SYNTAX scores. Nevertheless, in patients with a high SYNTAX score, a trend towards better survival was noted with CABG. The proportion of patients with a high SYNTAX score was limited in view of the inclusion criteria of the respective studies. Current evidence indicates that PCI is an appropriate alternative to CABG in LMCA and low-to-intermediate anatomical complexity. Among patients with LMCA and low anatomical complexity, there is evidence that the outcomes with respect to major clinical endpoints are similar for PCI and CABG, resulting in a class I recommendation. Among patients with LMCA and high anatomical complexity, the number of patients studied in RCTs is low due to exclusion criteria; the risk estimates and cIs are imprecise but suggest a trend towards better survival with CABG. Therefore, PCI in this setting cannot be endorsed as reflected by a class III recommendation. For PCI in LMCA with intermediate anatomical complexity, the previous class iIa recommendation was maintained in view of the incomplete 5-year follow-up of the two largest RCTs in this setting.
3. Percutaneous coronary intervention with drug-eluting stents for left main coronary artery disease

   The optimal DES therapy for patients with significant LMCA disease undergoing percutaneous coronary intervention (PCI) in contemporary practice remains undetermined. In the Intracoronary Stenting and Angiographic Results: Drug-Eluting Stents for Unprotected Coronary Left Main Lesions (ISAR-LEFT MAIN-2) (n=650) trial, the cumulative incidence of the primary endpoint, a composite of all-cause death, myocardial infarction, or target lesion revascularization was 17.5% in the thin-strut durable polymer zotarolimus-eluting stent group (Resolute, Medtronic, USA) and 14.3% in the thin-strut biocompatible durable polymer everolimus-eluting stent group (Xience®, Abbott Vascular, USA) (relative risk 1.26; 95% CI]: 0.85 to 1.85; p=0.25) at 12 months. In the Evaluation of XIENCE versus Coronary Artery Bypass Surgery for Effectiveness of Left Main Revascularization (EXCEL) trial, the rates of the primary composite endpoint of all-cause death, stroke, or MI, occurred similarly in patients undergoing PCI with the newer-generation thin-strut durable polymer everolimus-eluting stent (Xience®) and coronary artery bypass graft surgery (CABG) (22.0% vs. 19.2%, p=0.13) at 5 years. In the Nordic-Baltic-British left main revascularisation (NOBLE) trial, the rates of the primary composite endpoint of all-cause death, non-procedural MI, any repeat coronary revascularization, and stroke, was 29% in patients undergoing PCI with a thick-strut biodegradable polymer biolimus-eluting stent (Biomatrix Flex®, Biosensors, Switzerland) versus 19% in patients undergoing CABG (HR 1.48, 95% CI 1.11-1.96, CABG significantly better than PCI, p=0.0066) at 5 years. In the Improved Drug Eluting stent for All-comers Left Main (IDEAL-LM) randomized clinical trial, the rate of the primary endpoint, a composite of all-cause death, MI, or clinically indicated target vessel revascularization at 2 years did not differ between patients undergoing PCI with a biodegradable polymer everolimus-eluting stent (Synergy®, Boston Scientific, USA) combined with 4-month Dual Antiplatelet Therapy (DAPT) (14.6%) and those undergoing PCI with a durable polymer everolimus-eluting stent (Xience®, Abbott Vascular, USA) combined with 12-month DAPT (11.4%) (p=0.17). Newer-generation thin-strut polymer-free drug-coated stents have the potential to further mitigate chronic inflammation and promote faster re-endothelialisation. No dedicated randomized clinical trial to date has evaluated the safety and efficacy of newest-generation polymer-free drug-coated stents for PCI in patients with LMCA disease.
4. Antiplatelet therapy after percutaneous coronary intervention for left main coronary artery disease

   The 2018 ESC guidelines on myocardial revascularization recommend at least 6 (chronic coronary syndrome) and 12 (acute coronary syndrome) months of DAPT after PCI with newer-generation DES among patients with unprotected LMCA stenosis. However, a recent meta-analysis of five large-scale randomized clinical trials including a total of 32'145 patients, of whom 972 (3%) patients were treated for LMCA disease, indicated that 1-3 months of DAPT followed by P2Y12 inhibitor single antiplatelet therapy (SAPT) after second-generation DES implantation in patients with chronic and acute coronary syndromes was associated with lower risk for major bleeding (random-effects model: HR 0.63, 95% 0.45-0.86) and similar risk for stent thrombosis (random-effects model: HR 1.19, 95% CI 0.86-1.65), all-cause death (random-effects model: HR 0.85, 95% CI 0.70-1.03), MI (random-effects model: HR 1.05, 95% CI 0.89-1.23), and stroke (random-effects model: HR 1.08, 95% CI 0.68-1.74) compared with conventional DAPT. These findings suggest that a potent P2Y12 inhibitor-based SAPT following a short DAPT course (1-3 months) may represent a preferable treatment option, which is associated with similar ischemic, but lower bleeding risk, for patients undergoing PCI with newer-generation DES compared to standard conventional 12 months DAPT. However, the safety and efficacy of a potent P2Y12 receptor inhibitor-based aspirin-free SAPT after complex PCI, such as PCI for LMCA disease, has not been investigated to date.
5. Newer-generation ultrathin-strut drug-eluting stents for percutaneous coronary intervention

Newer-generation drug-eluting stents with ultrathin-strut metallic platforms have been shown to reduce the risk of target lesion failure compared with thicker-strut drug-eluting stents among all-comer patients undergoing PCI, a difference mainly driven by a lower risk of ischemia-driven target lesion revascularization. Supraflex Cruz (Sahajanand Medical Technologies Ltd., Surat, India) is a novel newer-generation drug-eluting stent consisting of an L-605 cobalt-chromium alloy metallic stent platform with ultrathin struts (60 μm) across all stent diameters, highly flexible S-link connectors, and a biodegradable polymeric matrix coating (poly L-lactide, 50:50 mixture poly D,L-lactide-co-glycolide and polyvinyl pyrrolidone) eluting sirolimus at a concentration of 1.4 μg/mm2 which is coated on the conformal surface of the stent together with the polymeric matrix. The average thickness of coating ranges from 4 to 5 μm. The drug is 70% released within 7 days, and the remainder is released over a period of 48 days. The polymer gradually degrades over 9-12 months. The proprietary 'LDZ' link design improves stent flexibility, transmits push force with higher efficiency, improves overall radial strength, and resists longitudinal compression. The open-cell design allows for better flexibility and facilitates side branch access. In addition, the 4.0 and 4.5 mm 8-crown stent platforms which allow for an overexpansion capacity up to 5.5 mm facilitates the treatment of patients with large coronary vessels, such as those undergoing LM PCI. In the TALENT prospective, single-blind, multicenter, randomized controlled trial that included 1'435 all-comer patients undergoing PCI, the Supraflex ultrathin-strut biodegradable polymer sirolimus-eluting stent was found non-inferior to the Xience® thin-strut permanent polymer everolimus-eluting stent (Abbott Vascular, USA) with regards to the device-oriented composite clinical endpoint (DoCE), a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization, at 12 months of follow-up. At 3 years, DoCE occurred in 57 patients (8.1%) in the Supraflex group, and in 66 patients (9.4%) in the XIENCE group (p=0.406). There were no significant between-group differences in rates of cardiac death, target vessel myocardial infarction or clinically indicated target lesion revascularization. The rates of definite or probable stent thrombosis were low and similar between groups (1.1% vs 1.4%; p=0.640). However, the TALENT trial included only 31 (1.5%) lesions located in the left main coronary artery and randomized evidence regarding the safety and efficacy of the Supraflex ultrathin-strut biodegradable polymer sirolimus-eluting stent for PCI in patients with significant LMCA disease remains therefore limited. The TAXCO study investigated the OCT-derived neointimal coverage of the Supraflex Cruz ultrathin-strut biodegradable polymer DES showing that 97.6% of the device struts are endothelialized at 6 months after PCI, which is comparable to the neointimal coverage of the Xience thin-strut everolimus-eluting stent. Equally, no significant difference was found with respect to 6months uncovered and malapposed struts between the 2 devices. Similarly, the SiBi study evaluated the early (4 to 6 weeks) OCT-derived neointimal coverage of the Supraflex Cruz ultrathin-strut biodegradable polymer DES demonstrating an excellent healing profile with a mean of 91.26% strut coverage at 35.3 ± 5 days after the index PCI. Taken together these results indicate an appropriate balance between neointimal thickness and amount of strut coverage that may facilitate short DAPT durations. Particularly, the use of thin strut and ultrathin strut stents may lead to a favorable trade-off in bleeding and ischemic events in patients with high-bleeding risk. In the COMPARE 60/80 HBR investigator-initiated, multicenter, prospective randomized trial which included a total of 732 patients at high-bleeding risk undergoing PCI with the Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent or the Ultimaster Tansei (Terumo Corp., Tokyo, Japan), the rates of the primary endpoint of the net adverse clinical endpoint, defined as a composite of cardiac death, myocardial infarction, target vessel revascularization, stroke, or BARC 3 or 5 major bleeding events at 12 months were 15.4% in the Supraflex Cruz group and 17.1% in the Ultimaster Tansei group, meeting the prespecified criterion for non-inferiority of the Supraflex Cruz DES compared to the Ultimaster Tansei DES (p=0.02). The median DAPT duration was 30 (0-181) days. Importantly, a lower rate of target lesion revascularization was observed in the Supraflex Cruz group in comparison to the Ultimaster Tansei group (2.7% vs. 5.3%, p=0.078). Additionally, most other cardiac endpoints showed numerically lower values in the Supraflex Cruz group when compared to the Ultimaster Tansei group. The safety and efficacy of the Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India) combined with potent P2Y12 inhibitor aspirin-free SAPT among all-comer patients undergoing PCI for complex coronary lesions, such as patients with LMCA stenosis, have however not been investigated to date.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patient with chronic or acute coronary syndrome (unstable angina, or non-ST-elevation acute coronary syndrome).
* Subject with significant unprotected (ostial, mid-shaft, or distal) LMCA stenosis who underwent successful LMCA PCI with ≥1 Supraflex Cruz ultrathin-strut biodegradable polymer sirolimus-eluting stent (Sahajanand Medical Technologies Ltd., Surat, India) according to current ESC guidelines on myocardial revascularization and/or local Heart Team decision.
* Subject willing to participate and able to understand, read and sign the informed consent document before the planned procedure.

Exclusion Criteria:

* Contraindications to PCI and/or DES implantation.
* Inability to adhere to DAPT for at least 6 months.
* Patient already on DAPT.
* Patients on oral anticoagulation.
* Previous coronary artery bypass surgery.
* LMCA in-stent restenosis or stent thrombosis.
* Recent ST-elevation myocardial infarction <5 days prior to randomization.
* Cardiogenic shock/hemodynamic instability at the time of intervention and/or need for mechanical/pharmacologic hemodynamic support.
* Participation or planned participation in another clinical trial, except for observational registries.
* Life expectancy <1 year.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite endpoint (POCE) | 2 years
  Composite of all-cause death, any non-fatal myocardial infarction, or any revascularization (PCI, or CABG)

SECONDARY OUTCOMES:
Net adverse clinical and major adverse cardiac (NACE) | 2 years
  Composite of all-cause death, any non-fatal myocardial infarction, any revascularization (PCI, or CABG), or Bleeding Academic Research Consortium (BARC)19 3 or 5 major bleeding
Device-oriented composite endpoint (DOCE) | 2 years
  Composite of cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization (PCI, or CABG)
All-cause death | 2 years
  Cardiac and non-cardiac death
Any non-fatal myocardial infarction | 2 years
  Periprocedural or spontaneous, target vessel-related, and non-target vessel-related myocardial infarction
Any revascularization | 2 years
  Any revascularization (PCI or CABG)
Target lesion revascularization | 2 years
  Clinically indicated and non-clinically indicated target lesion revascularization
Clinically indicated target vessel revascularization | 2 years
  Clinically indicated and non-clinically indicated target vessel revascularization
Definite stent thrombosis | 2 years
  Academic Research Consortium definite stent thrombosis
Definite or probable stent thrombosis | 2 years
  Academic Research Consortium definite or probable stent thrombosis
Bleeding Academic Research Consortium 3 or 5 major bleeding events | 2 years
  BARC 3 or 5 major bleeding complications
Bleeding Academic Research Consortium ≥2 major bleeding events | 2 years
  BARC ≥2 major bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Iglesias, MD, Principal Investigator — Geneva University Hospitals, Switzerland
Locations (1):
- Zurich University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request to the principal investigator after publication of the study primary and secondary endpoints.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study primary and secondary endpoints.